CLINICAL TRIAL: NCT07160049
Title: Focused Ultrasound Stimulation of Peripheral Nerves in Limbs
Brief Title: Wearable Focused Ultrasound Stimulation for Peripheral Nerve Pain Management
Acronym: PERNEUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Evan (Huiliang) Wang, Assistant Professor, University of Texas at Austin
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: STUDY00005942
Record Dates: First submitted 2025-07-25; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Pain Management; Peripheral Neuropathic Pain
Keywords: Focused Ultrasound; Peripheral Nerve Stimulation; Wearable Neurotechnology; Non-Invasive Neuromodulation; Pain Threshold; Pain Modulation; Radial Nerve; Tibial Nerve; Saphenous Nerve; Experimental Pain Testing; Ultrasound Neuromodulation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: This study uses a within-subject crossover design in which each participant completes nine sessions on separate days (~1 hour each). For each task (cold pressor, upper limb algometry, lower limb algometry), participants undergo three conditions: baseline assessment, sham stimulation, and active FUS stimulation. Sessions are scheduled on separate days to avoid carryover effects. Each participant serves as their own control, allowing direct comparison of responses to sham and active conditions.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Focused Ultrasound (FUS) Stimulation (Experimental): Participants will receive active focused ultrasound stimulation applied to peripheral nerves (radial, median, ulnar, tibial, saphenous, or peroneal) using a wearable FUS device. Stimulation will be performed during pain sensitivity assessments, including cold pressor tests and pressure algometry, to record pain perception/thresholds as exploratory physiological responses during feasibility testing.
  Interventions: Device: Cold Pressor Task - Upper Limb; Device: Algometry Pain Tests in the Upper Limb; Device: Algometry Pain Tests in the Lower Limb
- Sham Focused Ultrasound (FUS) Stimulation (Sham Comparator): Participants will undergo the same procedures as the experimental arm (device placement, cold pressor test, and pressure algometry) but with the FUS device set to sham (no active ultrasound output). This arm is used to control for placebo and non-specific effects of device application during pain sensitivity assessments.
  Interventions: Device: Cold Pressor Task - Upper Limb; Device: Algometry Pain Tests in the Upper Limb; Device: Algometry Pain Tests in the Lower Limb

INTERVENTIONS:
Device: Cold Pressor Task - Upper Limb — This study uses a three-session cold pressor paradigm to evaluate feasibility of a wearable focused ultrasound (FUS) device for peripheral nerve stimulation.
  Session 1 (Baseline): After consent, participants immerse the dominant hand in 0-1 °C water (~10 cm depth) in an insulated bucket. Time to first pain is recorded, with 5 min rests between immersions (12 total; max single immersion 6 min). Water temperature is digitally monitored, with ice added as needed.
  Session 2 (Sham): The median/ulnar/radial nerve in the dominant forearm is located by ultrasound. The FUS device is applied with hydrogel but set to sham (no output). The cold pressor protocol is repeated.
  Session 3 (Active FUS): After nerve localization, active FUS (650 kHz, 60-100% intensity, 20-30% duty cycle) is delivered for 5 min. The cold pressor test is repeated to record pain tolerance as an exploratory physiological response during feasibility testing.
Device: Algometry Pain Tests in the Upper Limb — This session records pressure pain thresholds in the dominant hand with a wearable FUS device and a pressure algometer during feasibility testing.
  Session 1 (Baseline): After consent and briefing, the median, ulnar, and radial nerves at three points on the dominant hand (wrist, palm, finger) are located via ultrasound and marked. A pressure algometer is applied to each site, with pressure gradually increased until pain is first reported. Thresholds are recorded, with each location tested three times with short breaks.
  Session 2 (Sham): The same nerve sites are identified and marked. The wearable FUS device is applied with hydrogel but set to sham (no active output). The baseline algometry protocol is repeated.
  Session 3 (Active FUS): Following nerve localization, active FUS (650 kHz, 60-100% intensity, 20-30% duty cycle) is delivered for 5 min. The algometry test is repeated to record pressure pain thresholds as exploratory physiological responses during feasibility testing.
Device: Algometry Pain Tests in the Lower Limb — This session records pressure pain thresholds in the dominant foot with a wearable FUS device and a pressure algometer during feasibility testing.
  Session 1 (Baseline): After consent and briefing, the tibial, saphenous, and peroneal nerves at three standardized points on the dominant foot are located via ultrasound and marked. A pressure algometer is applied to each site, and pressure is gradually increased until pain is first reported. Thresholds are recorded, with repeated trials and short breaks between tests.
  Session 2 (Sham): The same nerve sites are identified and marked. The wearable FUS device is applied with hydrogel but set to sham (no active output). The baseline algometry protocol is repeated.
  Session 3 (Active FUS): Following nerve localization, active FUS (650 kHz, 60-100% intensity, 20-30% duty cycle) is delivered for 5 min. The algometry test is then repeated to record pressure pain thresholds as exploratory physiological responses during feasibility testing.

SUMMARY:
This study will evaluate the feasibility of a novel wearable focused ultrasound (FUS) device for peripheral nerve stimulation in healthy volunteers. The aim is to assess device operability, usability, tolerability, and physiological responses during standardized sensory tests. Each participant will complete nine ~1-hour study sessions across multiple days, including cold pressor and algometry tasks performed under baseline, sham, and active FUS conditions.

DETAILED DESCRIPTION:
This feasibility study will evaluate a wearable focused ultrasound (FUS) system designed for non-invasive peripheral nerve stimulation of upper and lower extremity nerves. The primary objective is to determine device feasibility - operability, tolerability, usability, and physiological responses - during standardized pain sensitivity tasks.

Each participant will complete nine sessions on separate days (~1 hour each) in a within-subject crossover design:

1. Cold pressor test (baseline, sham, active FUS) - 3 days
2. Upper limb algometry (baseline, sham, active FUS) - 3 days
3. Lower limb algometry (baseline, sham, active FUS) - 3 days

Sessions will be scheduled at least 24 hours apart to avoid carryover effects. Approximately 12-15 participants will be enrolled. Although feasibility studies often include fewer than 10 participants, this sample size was chosen to ensure variability across limb anatomy and usability testing. No efficacy hypotheses or clinical outcomes will be tested.

ELIGIBILITY:
Inclusion Criteria:

- Healthy adults aged 20-40, willing and able to undergo FUS experiments.

Exclusion Criteria:

* Major physical illnesses.
* Diagnosis of a cognitive disorder.
* Cardiovascular conditions (e.g., high blood pressure, heart disease, or dysrhythmia), history of fainting or seizures, or history of frostbite.
* Open cuts, sores, or bone fractures on the limb to be immersed in water, or a history of Raynaud's phenomenon.
* Diagnosis of hypersensitivity or hyposensitivity to bodily sensations (temperature, vibrotactile, nociception).
* Inability to provide informed consent for FUS stimulation.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Completion Rate of Study Sessions | Through study completion (9 study visits over approximately 3 weeks).
  Proportion of participants who complete all nine planned sessions (baseline, sham, active FUS for cold pressor, upper limb algometry, and lower limb algometry) without withdrawal or device malfunction.

SECONDARY OUTCOMES:
Cold Pressor Pain Onset Time | 3 separate study visits (~1 hour each) over approximately 1 week.
  Time (seconds) from immersion of the hand in ice water until pain is first reported; measured during baseline, sham, and active FUS sessions to characterize physiological response during feasibility testing (not powered for efficacy).
Upper Limb Algometry Pain Threshold | 3 separate study visits (~1 hour each) over approximately 1 week.
  Maximum tolerated pressure (kgf) at standardized points on the hand and forearm before pain is reported, measured using a pressure algometer during baseline, sham, and active FUS sessions. Recorded as an exploratory physiological response during feasibility testing.
Lower Limb Algometry Pain Threshold | 3 separate study visits (~1 hour each) over approximately 1 week.
  Maximum tolerated pressure (kgf) at standardized points on the foot before pain is reported, measured using a pressure algometer during baseline, sham, and active FUS sessions. Recorded as an exploratory physiological response during feasibility testing.

CONTACTS AND LOCATIONS:
Overall Officials: Huiliang Wang, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Biomedical Enginering Building - UT Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lotz G, Stahlschmidt M. [Agenesis of the gallbladder]. Chirurg. 1986 Jan;57(1):37-9. No abstract available. German. PMID 3514181
- [Background] Patrini C, Reggiani C, Laforenza U, Rindi G. Effect of acute and chronic ethanol administration on the transport of thiamine from plasma to different brain regions of the rat. Alcohol Alcohol. 1988;23(6):455-63. PMID 3245865